CLINICAL TRIAL: NCT03718754
Title: En-bloc vs Conventional Resection of Primary Bladder Tumor: Prospective Randomized Multicenter Trial
Brief Title: En-bloc vs Conventional Resection of Primary Bladder Tumor
Acronym: eBLOC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: David D'Andrea (Other)
Responsible Party: Sponsor-Investigator, David D'Andrea, M.D., Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1636/2018
Record Dates: First submitted 2018-10-23; First posted 2018-10-24 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- En-Bloc TURB (Active Comparator)
  Interventions: Device: En-Bloc TURB
- Conventional TURB (Active Comparator)
  Interventions: Device: Conventional TURB

INTERVENTIONS:
Device: En-Bloc TURB — En-bloc resection will be performed at each center based on local clinical practice and available instruments. Laser resection, hydrodissection with HybridKnife® or electric resection are allowed. All procedures, including cTURB, must be performed with an imaging enhancing technique (PDD / NBI at surgeon's discretion). After resection, a single intravesical instillation of 40mg Mitomycin-C will be performed if clinically feasible.
  Arms: En-Bloc TURB
Device: Conventional TURB — En-bloc resection will be performed at each center based on local clinical practice and available instruments. After resection, a single intravesical instillation of 40mg Mitomycin-C will be performed if clinically feasible.
  Arms: Conventional TURB

SUMMARY:
Based on current evidence, we hypothesize that eTURB represents an improvement in the surgical management of NMIBC. The resection is more precise and complete compared to cTURB. Moreover, the quality of an en-bloc specimen, including the tumor with its adjacent bladder wall layers, allows an accurate pathological review which leads to correct risk allocation and therapy.

To answer these questions, we designed a RCT comparing eTURB with cTURB. Primary outcome of our study will be the accuracy of pathological staging assessment measured by the presence of detrusor muscle in the specimen as a surrogate parameter for quality of resection.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet all the following inclusion criteria to participate in this study:

* Diagnosis by cystoscopy of primary papillary non-muscle invasive bladder urothelial carcinoma (cTa, cT1)
* Imaging examinations shows that the bladder muscle has not been affected, no lymph node metastasis or distant metastasis;
* Diameter of tumor between 1cm and 3cm
* Number of lesions ≤3 (The position of small lesions relatively concentrated as one place)
* Patients who agree to eTURB or cTURB surgery, and will be effected to the postoperative follow-up treatment such as conventional infusion after the operation

Exclusion Criteria

* Pure carcinoma in situ
* Contraindications to surgery (i.e. bladder fibrosis)
* Diameter of tumor >3cm
* Number of lesions >3
* Poor performance status making a surgical intervention too risky
* Life expectancy of less than one year
* Patient refused to participate
* Pregnancy
* History of upper urinary tract malignancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
The pathological staging assessment for eTURB compared to cTURB | 4 weeks
  The primary objective of the study is to assess whether eBLOC is associated with a higher rate of detrusor muscle in the pathologic specimen, compared to cTURB

SECONDARY OUTCOMES:
Residual disease within 3 months after initial TURB | 3 months
Occurrence of obturator reflex | 1 day
Operative time | 1 day
Number of participants with bladder perforation | 7 days
Upstaging of disease upon second look transurethral resection surgery | 6 weeks
Number of participants with obturator reflex | 1 day
Number of tumors with evaluable lateral and deep resection margin | 4 weeks
Number of tumors with positive lateral and deep resection margin | 4 weeks
Number of participants with conversion to other resection technique | 1 day
Number of participants with persistent disease at 2nd look TURB | 6 weeks
Recurrence-free survival | up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Shahrokh Shariat, M.D., Study Chair — Shahrokh.shariat@meduniwien.ac.at
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] D'Andrea D, Soria F, Hurle R, Enikeev D, Kotov S, Regnier S, Xylinas E, Lusuardi L, Heidenreich A, Cai C, Frego N, Taraktin M, Ryabov M, Gontero P, Comperat E, Shariat SF; eBLOC Study Team. En Bloc Versus Conventional Resection of Primary Bladder Tumor (eBLOC): A Prospective, Multicenter, Open-label, Phase 3 Randomized Controlled Trial. Eur Urol Oncol. 2023 Oct;6(5):508-515. doi: 10.1016/j.euo.2023.07.010. Epub 2023 Aug 4. PMID 37543464